CLINICAL TRIAL: NCT05891002
Title: Diagnostic Accuracy of Robotically Assisted Cranial Biopsies Using Cirq Active Cranial and Automatic Image Registration
Brief Title: Accuracy of Robotically Assisted Cranial Biopsies
Status: Recruiting | Type: Observational
Sponsor: Brainlab AG (Industry)
Responsible Party: Sponsor
Other Study IDs: Angers-Cirq Cranial-01
Record Dates: First submitted 2023-05-26; First posted 2023-06-06 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Intracranial Neoplasm
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Biopsy Patient: Patient with a confirmed intracranial neoplasm scheduled for a biopsy with Cirq® Robotic Alignment Module Cranial and registration via Auto-Registration Software Universal Automatic Image Registration Cranial and Loop-X® Mobile Imaging Robot.
  Interventions: Device: Cirq® Robotic Alignment Module Cranial

INTERVENTIONS:
Device: Cirq® Robotic Alignment Module Cranial — Robotic navigation for cranial biopsy procedure

SUMMARY:
This is an observational post-market study determining biopsy accuracy in a clinical environment using Cirq® Robotic Alignment Module Cranial. The goal is to determine whether the robotic procedure to be examined can achieve a clinically acceptable value of at least 90% in terms of diagnostic yield.

DETAILED DESCRIPTION:
The goals of the project are to determine the accuracy of Cirq® Robotic Alignment Module Cranial navigated biopsy procedures, Automatic Image Registration accuracy within the workflow, and compatibility of Cirq® Robotic Alignment Module Cranial in the clinical workflow. Patients will undergo cranial biopsies according to standard of care using released products within their intended use with the exception that the accuracy of the biopsy needle will be measured using a specific intraoperative workflow.

ELIGIBILITY:
Inclusion Criteria:

* Intracranial lesion and the indication for a diagnostic stereotactic biopsy validated by the neurosurgical staff
* Ability to consent to the procedure

Exclusion Criteria:

* Pregnancy
* Contraindications on narcosis, operation, CT scan, MRI scan and/or Gadolinium contrast agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 consecutive patients who are planned to undergo a brain biopsy will be included. Since this is a confirmatory study, a sample size calculation was not able to be performed.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | 24 months
  Determine the percentage of diagnostically significant biopsies determined histologically

SECONDARY OUTCOMES:
Target point and entry point error | 24 months
  Determine accuracy of biopsy needle by comparing the target and entry point location to the planned location
Time for procedure | 24 months
  Determine the time needed for the intraoperative biopsy procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Lemée, MD, Study Director — University Hospital, Angers
Locations (1):
- The Centre Hospitalier Universitaire (CHU) d'Angers health establishment, Angers, France